CLINICAL TRIAL: NCT04719962
Title: Diagnosis of Disseminated Lyme Borreliosis by Targeted Proteomics
Brief Title: Direct Diagnosis of Disseminated Lyme Borreliosis.
Acronym: DIALYD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7609
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Lyme Disease
Keywords: targeted proteomics; skin biopsy; biomarker
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disseminated Lyme infection (Experimental): Only patients presenting with disseminated Lyme borreliosis will be part of the study.
  Interventions: Procedure: Targeted proteomics in skin +/- cerebrospinal or synovial fluid to diagnose disseminated Lyme disease

INTERVENTIONS:
Procedure: Targeted proteomics in skin +/- cerebrospinal or synovial fluid to diagnose disseminated Lyme disease — Following a 2-days course of local daily clobetasol propionate 0,05% cream application, a skin biopsy (3 mm punch-biopsy ) of healthy-looking skin of the upper part of the thigh will be performed in all patients,.
  Arthrocentesis (in patients with Lyme arthritis only) and lumbar puncture to collect cerebrospinal fluid (in patients with neuroborreliosis only) will be performed in the usual care setting as appropriated.
  All biological samples will be subject to Borrelia culture, PCR and SRM-MS proteomics.

SUMMARY:
Lyme borreliosis is a bacterial multisystemic infection transmitted by an Ixodes tick. It affects the skin, the joint and the brain. At the early phase, the diagnosis is clinical, relying on the presence of an erythema migrans at the site of the tick bite. The diagnosis of disseminated infections, more difficult to assess, mainly relies on indirect diagnosis test, i.e. serology.

This study will evaluate a new direct diagnosis method based on proteomics, which aims to demonstrate proteins of live bacteria in the skin and the synovial or cerebrospinal fluids in a direct manner.

DETAILED DESCRIPTION:
Lyme borreliosis is a multisystemic bacterial infection affecting the skin, the joint and the nervous system. It has been shown that the skin is an essential interface as a site of bacteria inoculation and multiplication. In mouse acutely infected with different Borrelia species, the investigators have detected several protein markers of active infection in the skin by discovery proteomics, which allowed us to design a subsequent targeted proteomics assay. The invcestigators tested the same techniques in skin biopsies of humans presenting with an erythema migrans. Most of the bacterial proteins previously identified in the skin of infected mice were also detected in biopsies of human lesional skin.

The diagnosis of disseminated Lyme borreliosis currently mainly relies on evocative clinical symptoms along with a positive Borrelia serology. However, a positive serological test does not prove an active infection but merely reflects exposure to the pathogen, which is quite common in endemic regions and thus lacks positive predictive value. Moreover, direct bacteriological diagnosis tools such as culture and nucleic acid amplification (PCR) currently lack sensitivity. Planning to test the ability of proteomics to assist in the diagnosis of disseminated Lyme borreliosis, we have first developed a model of late infection in mouse, and achieved the identification of several bacterial proteins as markers of ongoing infection in the murine skin.

The investigators now wish to investigate whether the skin also constitutes a reservoir for these bacteria during persistent disseminated infection in humans, and if they can detect bacterial proteins in this easily accessible tissue by the same approach. They will directly look for bacterial proteins by selected reaction monitoring-mass spectrometry (SRM-MS), the method successfully employed in early infection setting. The ability to detect borrelial proteins in synovial fluid (patients with Lyme arthritis), cerebrospinal fluid (patients with Lyme neuroborreliosis) or lesional skin (patients with acrodermatitis chronica atrophicans) will also be investigated, as appropriated.

To improve the detection of Borrelia proteins in healthy-looking skin, a dermocorticoid will be prealably applied for a short 2-days course, a procedure the investigators demonstrated both useful and safe in mice. Since tick bite mainly occurs in the lower part of the body, the upper part of the thigh will be the site of topical steroids application and skin biopsy .

The proteomics yield will be compared to the two main other methods of direct detection, i.e. culture and PCR.

ELIGIBILITY:
Inclusion criteria:

* Subject over 18 years of age
* Subject informed of the results of the previous medical examination and informed about research objectives and risks
* Subject affiliated to a social health insurance
* Subject having signed informed consent
* Subject with clinical and serological criteria that meet the criteria of French societies, published in May and June 2019 (Jaulhac et al., 2019) as well as the European criteria of ESGBOR, corresponding to a disseminated infection of Lyme borreliosis.

Clinical Criteria:

* acute or subacute meningoradiculitis in a subject exposed to tick bites
* Uni- or bilateral peripheral facial paralysis in a subject exposed to tick bites
* Chronic radiculitis table compatible with Lyme borreliosis
* mono- or oligo arthritis of large jointsin the absence of other obvious diagnosis (inflammatory rheumatism flares, microcrystalline arthritis…)
* Skin changes suggestive of acrodermatitis chronica atrophicans

Serological criteria: positivity for Lyme serology (two-tiered, IgG)

Exclusion criteria:

* contraindication to performing a skin biopsy
* contraindication to local lidocaine anaesthesia with or without adrenaline
* contraindication to dermocorticoids (hypersensitivity)
* antibiotic treatment for borreliosis already administered
* inability to provide informed information
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2022-07-07 (Estimated)

PRIMARY OUTCOMES:
Direct diagnosis of disseminated Lyme disease by proteomics | 6 months
  1. Detection or not of targeted proteins by SRM-MS in healthy-looking skin samples of patients with disseminated Lyme borreliosis (either clinical presentation)
  2. Detection or not of targeted borrelial proteins by SRM-MS in synovial fluid of patients with Lyme arthritis
  3. Detection or not of targeted borrelial proteins by SRM-MS incerebrospinal fluid of patients with neuroborreliosis
  4. Detection or not of targeted borrelial proteins by SRM-MS in lesional skin of patients with acrodermatitis chronica atrophicans

CONTACTS AND LOCATIONS:
Overall Officials: Benoît JAULHAC, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided